CLINICAL TRIAL: NCT01743378
Title: Ultrasound Guided Transversus Abdominis Plane Block With Ropivacaine vs Placebo for Abdominal Hysterectomy: a Double-blinded, Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Billy B Kristensen, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1-2010-068
Record Dates: First submitted 2012-11-13; First posted 2012-12-06 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Pain and Postoperative Morphine Consumption After Abdominal Hysterectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP Block Ropivacaine 0,75 % (Experimental): Bilateral Transversus Abdominis Plane Block with 2 x 20 ml Ropivacaine 0,75 %
  Interventions: Procedure: TAP Block Ropivacaine 0,75 %
- TAP Block Saline 0,9 % (Placebo Comparator): Bilateral Transversus abdominis plane block with 2 x 20 ml Saline 0,9 %
  Interventions: Procedure: TAP Block Saline 0,9 %

INTERVENTIONS:
Procedure: TAP Block Ropivacaine 0,75 %
  Arms: TAP Block Ropivacaine 0,75 %
Procedure: TAP Block Saline 0,9 %
  Arms: TAP Block Saline 0,9 %

SUMMARY:
A Prospective double-blinded randomized clinical trial to test the effect of transversus abdominis plane block on postoperative pain and opoid consumption after abdominal hysterectomy.

Two groups of each 24 patients. All patients are given general anesthesia. The patients are randomized to have a ultrasound guided bilateral transversus abdominis plane block with either 2 x 20 ml 0,75 % ropivacaine or 2 x 20 ml of 0,9 saline. All patients are provided with a PCA for self administration of morphine.

Pain score on visual analog scale, nausea and vomiting are monitored at 1, 2, 4, 6, 8 and 24 hours postoperatively as well as the total consumption of morphine after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Assigned to elective abdominal hysterectomy
* Must be able to understand and speak danish
* Must be able to give verbal and written consent

Exclusion Criteria:

* Abuse of alcohol or medicin
* Daily treatment with opoids or glucocorticoids
* Allergy towards any kind of localanesthetic drug
* Intolerance toward morphine
* Psychiatric desease
* Age below 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption during first 24 hours postoperatively | At 24 hours postoperatively

SECONDARY OUTCOMES:
Postoperative pain by visual analog scale at | Monitored at 1, 2, 4, 6, 8 and 24 hours postoperatively
  Monitored at 1, 2, 4, 6, 8 and 24 hours postoperatively by one of the investigators at rest, when coughing and when walking

OTHER OUTCOMES:
Postoperative nausea and vomiting | Monitored at 1, 2, 4, 6, 8 and 24 hours postoperatively
  Monitored at 1, 2, 4, 6, 8 and 24 hours postoperatively by one of the investigators
Length of stay | First 72 hours after surgery
  Length of hospital stay counted in days
Time until mobilization | First 24 hours postoperatively
  First mobilization defined as walking on the floor

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Capital Region, Denmark